CLINICAL TRIAL: NCT00561782
Title: MR Spectroscopy (MRS) as a Diagnostic and Outcome Measure in Pain and SCI
Brief Title: MR Spectroscopy as a Diagnostic and Outcome Measure in Pain and SCI
Acronym: MRS
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of Miami (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: B5023-R
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Spinal Cord Injury; Hyperalgesia, Secondary; Hyperalgesic Sensations
Keywords: Spinal Cord Injury Pain; Chronic Neuropathic Pain; SCI Pain; Pain, Chronic Neuropathic; Spectroscopy, Magnetic Resonance; MRS; Traumatic Brain Injury Pain
MeSH Terms: conditions — Spinal Cord Injuries; Hyperalgesia; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group 1: Spinal cord injured with chronic central neuropathic pain.
- Group 2: Spinal cord injured without chronic central neuropathic pain.
- Group 3: Able-bodied without history of chronic pain of any type
- Group 4: Traumatically Brain Injured with a history of pain that onset after their TBI

SUMMARY:
The goal of this study is to compare the changes that occur in sensation and chemical properties of the brain following SCI between individuals that experience chronic pain and those that do not, and between those with SCI and the able-bodied.

DETAILED DESCRIPTION:
This study investigates the differences in certain neurochemicals present in areas of the brain linked to pain processing in people with SCI and neuropathic pain, in people with SCI but no pain, and in able-bodied persons. We will also investigate the relationship between these concentrations of neurochemicals and different aspects of chronic neuropathic pain, including the intensity of pain, quality of life issues, sensitivity changes in areas of the body that are both painful and non-painful, and neurological status.

ELIGIBILITY:
Inclusion Criteria:

1. SCI and neuropathic pain:

   * fluent in English
   * incomplete or complete traumatic SCI
   * the injury must have occurred at least 2 years prior to entering the study
   * the injury level must be above L1 and the subjects must have evidence of preserved distal cord functions (lower extremity reflexes and bulbocavernosus or anal wink reflexes)
   * must have experienced chronic neuropathic pain at or below the level of injury for a minimum of six months
   * must have moderately severe or greater neuropathic pain
   * must be able to attend three sessions ranging from 2 to 6 hours over a period of 4 to 5 weeks
2. SCI and no neuropathic pain:

   - same as a., but participants in this group must NOT have unremitting moderate-severe pain and there will only be two sessions ranging from 2 to 6 hours over a period of 1 to 2 weeks
3. Able-bodied control subjects:

   * fluent in English
   * no history of chronic pain conditions
   * no substantial brain or body injury
   * must be able to attend two sessions ranging from 2 to 6 hours over a period of 1 to 2 weeks

Exclusion Criteria:

* current pregnancy or women who are contemplating pregnancy
* recent (one-year) history of alcohol or drug abuse
* known intra-cerebral pathology or epilepsy
* MRI findings indicative of intra-cerebral pathology
* significant post-traumatic encephalopathy from head trauma sustained at SCI or cognitive impairment indicative of traumatic brain injury
* current diagnosis of DSM-IV Axis I disorder
* inability to meet the MRI screening requirements (including, but not limited to, the presence of a pacemaker or other electronic devices, prosthesis, artificial limb or joint, shunt, some metal rods, some tattoos, or moderate to severe claustrophobia or anxiety)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both spinal cord injured (85) and able-bodied (25) subjects will be studied. Of those with spinal cord injury, 60 will be those who experience central neuropathic pain and 25 will not. An additional 25 people who screen positive for mild to moderate TBI symptoms and pain attributable to TBI will be studied.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2007-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Using MR Spectroscopy to measure the concentration of N-acetyl aspartate, glutamate/glutamine, and myo-inositol in the areas of the brain thought to process pain. | Two measures at intervals of 2 to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eva G. Widerstrom-Noga, DDS PhD, Principal Investigator — VA Medical Center, Miami
Locations (1):
- VA Medical Center, Miami, Miami, Florida, United States

REFERENCES:
- [Background] Eaton MJ, Widerstrom-Noga E, Wolfe SQ. Subarachnoid Transplant of the Human Neuronal hNT2.19 Serotonergic Cell Line Attenuates Behavioral Hypersensitivity without Affecting Motor Dysfunction after Severe Contusive Spinal Cord Injury. Neurol Res Int. 2011;2011:891605. doi: 10.1155/2011/891605. Epub 2011 Jun 1. PMID 21799949
- [Result] Widerstrom-Noga E, Pattany PM, Cruz-Almeida Y, Felix ER, Perez S, Cardenas DD, Martinez-Arizala A. Metabolite concentrations in the anterior cingulate cortex predict high neuropathic pain impact after spinal cord injury. Pain. 2013 Feb;154(2):204-212. doi: 10.1016/j.pain.2012.07.022. Epub 2012 Nov 8. PMID 23141478
- [Result] Cruz-Almeida Y, Felix ER, Martinez-Arizala A, Widerstrom-Noga EG. Decreased spinothalamic and dorsal column medial lemniscus-mediated function is associated with neuropathic pain after spinal cord injury. J Neurotrauma. 2012 Nov 20;29(17):2706-15. doi: 10.1089/neu.2012.2343. Epub 2012 Aug 27. PMID 22845918
- [Result] Felix ER, Widerstrom-Noga EG. Reliability and validity of quantitative sensory testing in persons with spinal cord injury and neuropathic pain. J Rehabil Res Dev. 2009;46(1):69-83. PMID 19533521
- [Result] Cruz-Almeida Y, Alameda G, Widerstrom-Noga EG. Differentiation between pain-related interference and interference caused by the functional impairments of spinal cord injury. Spinal Cord. 2009 May;47(5):390-5. doi: 10.1038/sc.2008.150. Epub 2008 Nov 25. PMID 19030010
- [Result] Widerstrom-Noga EG, Cruz-Almeida Y, Felix ER, Adcock JP. Relationship between pain characteristics and pain adaptation type in persons with SCI. J Rehabil Res Dev. 2009;46(1):43-56. PMID 19533519